CLINICAL TRIAL: NCT02482688
Title: A Randomised Controlled Study of Early vs. Late, and Unisensory vs. Multisensory Rehabilitation for Stroke Patients With Perceptual and Cognitive Impairments.
Brief Title: A New Rehabilitation Treatment Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/SC/1339; 160140 (Other: Clinical trial CSP ref:)
Record Dates: First submitted 2015-06-23; First posted 2015-06-26 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multisensory Acute (Experimental): Multisensory intervention delivered within 2 months post-stroke.
  Interventions: Behavioral: A New Rehabilitation Treatment following Stroke
- Multisensory Chronic (Experimental): Multisensory intervention delivered 6 months post-stroke.
  Interventions: Behavioral: A New Rehabilitation Treatment following Stroke
- Unisensory Acute (Active Comparator): Unisensory intervention delivered within 2 months post-stroke.
  Interventions: Behavioral: A New Rehabilitation Treatment following Stroke
- Unisensory Chronic (Active Comparator): Unisensory intervention delivered 6 months post-stroke.
  Interventions: Behavioral: A New Rehabilitation Treatment following Stroke

INTERVENTIONS:
Behavioral: A New Rehabilitation Treatment following Stroke — A randomised control design, comparing individuals who will receive visual unisensory stimulation alone (i.e., the control rehabilitation) and those who receive multisensory stimulation (i.e., the experimental rehabilitation), will be used to assess the effects of multisensory rehabilitation on learning, performance accuracy and speed in participants with neglect/extinction.
  Other Names: A randomised controlled study of early vs. late, and unisensory vs. multisensory rehabilitation for stroke patients with perceptual and cognitive impairments.

SUMMARY:
Stroke is the number one cause of disability in the United Nations with about 1 million new cases each year. Following stroke, patients with perceptual and cognitive impairments have the worst prognostic outcomes. There is evidence to suggest that perceptual and cognitive symptoms can be alleviated by multisensory integration, which has the effect of enhancing motor, perceptual and cognitive processes. This research project will investigate for the first time the functional benefits that stem from multisensory stimulation of attention in stroke patients with perceptual and cognitive impairments. The research project will involve multisensory learning paradigms with stimulus and environmental parameters that optimally enhance perceptual learning and cognitive function. Multisensory learning paradigms will be tailored for patients with stroke to determine the perceptual and cognitive symptoms that can be alleviated, and fMRI will be used to evaluate the underlying neural substrates of the effects. The project will show whether multisensory stimulation provides an effective means of attentional rehabilitation after stroke and whether the effects generalize to everyday life, with long-term outcomes that improve functional independence in patients with stroke.

DETAILED DESCRIPTION:
Stroke is one of the major causes of death worldwide, second only to coronary disease, and it is the leading cause of disability with patients needing long hospitalisation and long-term community care (Mackay, Mensah, Mendin, & Greenlund, 2004). Stroke patients with perceptual and cognitive impairments such as unilateral neglect are of particular concern as they have among the worst prognostic outcomes (Di Monaco et al., 2011; Narasimhalu et al., 2011). Unilateral neglect, commonly observed after brain damage of the right posterior parietal cortex, is most often associated with reduced awareness of visual or auditory stimuli presented to the contralesional (left) side of space (Humphreys & Riddoch, 2001), particularly in the presence of competing stimuli on the ipsilesional (right) side (i.e., extinction) (Humphreys, Romani, Olson, Riddoch, & Duncan, 1994). This can manifest as a failure to cancel lines on one side of a page ('neglect'). In milder cases the patient can detect a single stimulus on the contralesional side but fails to detect the same item when another item is presented simultaneously on the ipsilesional side ('extinction'). Currently there is no consensus about optimal training strategies to alleviate neglect and extinction, therefore, it remains important to attempt to develop new procedures that are effective in the medium to long-term, that generalise outside the clinic and that are clinically applicable.

Multisensory integration is a potentially important vehicle for neurorehabilitation because it is known to generate large facilitative effects on information processing across a wide range of individuals. For example, motor reaction times (RTs) are significantly faster (Barutchu, Crewther, & Crewther, 2009; Barutchu, Freestone, Innes-Brown, Crewther, & Crewther, 2013), and perceptual sensitivities (Stein, London, Wilkinson, & Price, 1996), working memory and learning (e.g., Shams & Seitz, 2008), are enhanced in response to spatially and temporally synchronous multisensory stimuli when compared with stimuli presented in a single sensory modality. In addition, multisensory integration can be used to compensate for unisensory decline in the elderly by restoring motor function to levels generally observed in younger adults (e.g., Laurienti, Burdette, Maldjian, & Wallace, 2006). Critically, recent evidence suggests that some stroke patients in general may benefit from early post-stroke rehabilitation (Bai et al., 2012), and that some stroke patients with heminopia can benefit from multisensory integration (e.g., Passamonti, Bertini, & Ladavas, 2009). These studies have also demonstrated that multisensory rehabilitation strategies can have long lasting effects up to 1 year after initial training, and that improvements can generalize to other daily activities, such as reading. However, it is unknown whether these findings can be generalized to other types of perceptual and cognitive impairments. This study will be the first to investigate the combined long-term effects of multisensory signals and establish when is it more effective to intervene during the acute or chronic stage of the disorder.

The aim of this project is to develop a novel approach to the remediation of neglect and extinction by comparing multisensory integration with unisensory integration, and determining whether it is best to intervene during the acute or chronic stage of the disorder. In addition, the project will investigate the neural underpinning of functional recovery in neglect patients, using fMRI.

The specific aims of this research project are:

* To assess if perception can be improved in stroke patients with unilateral neglect/extinction as a result of multi- or uni-sensory integration, how well training effects generalize to other tasks and their longevity when the rehabilitation is delivered in the acute stage vs. the chronic stage of the disorder.
* To evaluate, using functional magnetic resonance imaging (fMRI), adaptive changes and plasticity in brain networks following multisensory learning in patients with neglect/extinction, so that an understanding is gained of the neural mechanisms linked to functional recovery in neglect/extinction patients.

Description of the rehabilitation

A randomised control design, comparing individuals who will receive visual unisensory stimulation alone (i.e., the control rehabilitation) and those who receive multisensory stimulation (i.e., the experimental rehabilitation), will be used to assess the effects of multisensory rehabilitation on learning, performance accuracy and speed in participants with neglect/extinction. Participants with neglect/extinction will be recruited between 2 days - 2 months post stroke and randomly allocated into one of 4 groups: 2 stages post-stroke (acute vs. chronic) x 2 rehabilitation types (unisensory vs. multisensory) (~20 participants per group). Search and memory tasks will be developed where participants are presented with only visual stimuli (e.g., objects - unisensory stimulation groups) or both visual stimuli and sounds (multisensory stimulation groups). Participants will be presented with the stimuli and asked to detect or remember the objects or their locations. Participant will have the option of responding verbally or by pressing a button. Task will begin at an easy level (e.g., one object being presented at a time) and gradually increase in difficulty as participant performance improves (e.g., by increasing the number objects to be detected or remembered). All participants will be subjected to 2 weeks of unisensory or multisensory rehabilitation (6 sessions approximately every second day). The rate of improvement across sessions will be measured in order to judge the best training 'dose' to use in future clinical settings. To gauge recovery, and its generalisation across other cognitive processes, and its long-term carry over effects, participants will be assessed using the Birmingham Cognitive Screen (BCoS) and the Oxford Cognitive Screen (OCS)(Humphreys, Bickerton, Samson, & Riddoch, 2012) before and at 1- and 6-months post rehabilitation. The investigators will also include measures of functional outcome (e.g., Stroke Impact Scale - SIS, and the Nottingham Extended ADL test) and measures of quality of life QoL (for the participant and carer).

At the beginning of the study (screening phase), all participants will be screened to assess their eligibility for the study and fMRI. Participants who meet the eligibility criteria will be invited to participate in the rehabilitation program (study phase). Only participants who meet the inclusion criteria for fMRI will be invited to have their brain scanned in study phase before the rehabilitation and 1-month post rehabilitation. For the fMRI scan, T1, Flair and DTI will be recorded and a simple detection task with auditory and visual stimuli will be used to measure functional activity to unilateral and bilateral stimulus presentations.

There are no known potential risks of the study, other than the well known contra-indication for MRI for participants who are invited to have their brain scanned, and the inconvenience of attending up to nine sessions: one at screening phase, six during the study phase, and two follow-up sessions at 1 month and 6 months following the completion of the 6th session in the study phase.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participants who have a history of stroke (within the last 2 days - 2 months) and demonstrate a clinical deficit in unilateral neglect and/ or extinction on our standardised measure from the Oxford Cognitive Screen (OCS) and/or extinction task from BCoS (Birmingham Cognitive Screen).
* Participants have sufficient comprehension and concentration to undergo cognitive screening lasting about 1 hour (BCoS sub-tests, and other neglect and extinction related tests).
* Participants are medically stable.
* Participants with no history of other neurological and psychiatric disorders with exception of stroke.

Exclusion Criteria:

* Participants unwilling or unable to give consent.
* Participants without cognitive deficits and unilateral neglect or extinction.
* Participants who cannot concentrate sufficiently to undergo the screening and/or who are not medically stable.
* Participants with a history of other neurological and psychiatric disorders (with exception of stroke).
* Counter-indicators for fMRI (only relevant to the brain scanning portion of the study). Participants with counter-indicators for fMRI will still be invited to take part in the rehabilitation program.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
The efficacy of multisensory vs. unisensory rehabilitation program for stroke participants with perceptual impairments at the acute vs. chronic stage of the disorder. | 4 years
  Changes in performance on neuropsychological tests throughout the rehabilitation program, and 1 month and 6 months post rehabilitation.

SECONDARY OUTCOMES:
Changes in brain networks related to the recovery of perceptual and cognitive functions. | 4 years
  Changes in neural network activity as assessed using fMRI and tractography at 1 month after the completion of the rehabilitation program compared with pre rehabilitation scans.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom